CLINICAL TRIAL: NCT07085273
Title: A Single-arm Clinical Study of Irinotecan Liposome II + 5-FU/LV + Oxaliplatin + Karelizumab for Neoadjuvant Treatment of Gastric Cancer
Brief Title: Irinotecan Liposome II + 5-FU/LV + Oxaliplatin + Karelizumab in Neoadjuvant Treatment of Gastric Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital of Zhengzhou University (Other)
Responsible Party: Principal Investigator, Yongxu Jia, Clinical Professor, The First Affiliated Hospital of Zhengzhou University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25-OBU-HN-GC-II-012
Record Dates: First submitted 2025-07-08; First posted 2025-07-25 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — irinotecan sucrosofate; Fluorouracil; Leucovorin; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Irinotecan liposomal+5-FU/Calcium folinate+Oxaliplatin+Karelizumab (Experimental): FOLFIRINOX + Karelizumab Irinotecan liposomal: 60 mg/m2, IV infusion, d1; 5-FU: 400 mg/m2, IV infusion, d1, followed by 1200 mg/m2/d x 2 days of continuous IV infusion (total 2400 mg/m2, 46-48h infusion); Calcium folinate: 400 mg/m2, IV infusion, d1; Oxaliplatin: 85 mg/m2, IV infusion, d1; Karelizumab: 200 mg, IV infusion, d1; Repeat every 2 weeks.
  Interventions: Drug: Irinotecan Liposomal

INTERVENTIONS:
Drug: Irinotecan Liposomal — FOLFIRINOX + Karelizumab Irinotecan liposomal: 60 mg/m2, IV infusion, d1; 5-FU: 400 mg/m2, IV infusion, d1, followed by 1200 mg/m2/d x 2 days of continuous IV infusion (total 2400 mg/m2, 46-48h infusion); Calcium folinate: 400 mg/m2, IV infusion, d1; Oxaliplatin: 85 mg/m2, IV infusion, d1; Karelizumab: 200 mg, IV infusion, d1; Repeat every 2 weeks.
  Other Names: 5-FU; Calcium folinate; Oxaliplatin; Karelizumab

SUMMARY:
For non-esophagogastric union progressive gastric cancer, the current treatment standard is D2 surgical resection combined with postoperative adjuvant chemotherapy, and for those with advanced stage (clinical stage III or above), perioperative chemotherapy mode can be chosen. For progressive esophagogastric combination cancer, neoadjuvant radiotherapy or preoperative chemotherapy can be chosen. Preoperative chemotherapy significantly improves the tumor remission rate and R0 resection rate with good safety. Irinotecan has been widely used in clinical practice, and together with the available data from the Irinotecan Liposome (II) clinical study demonstrated good safety and clinical efficacy, bringing hope for prolonging progression-free survival and overall survival for several tumor patients. In order to further explore the safety and efficacy of the neoadjuvant therapeutic application of irinotecan liposome (II) in patients with gastric cancer, the present study was conducted to provide data to guide future clinical practice.

ELIGIBILITY:
Inclusion Criteria:

1. age ≥ 18 years and ≤ 75 years;
2. gastric cancer confirmed by histopathology or cytology;
3. critically resectable gastric cancer confirmed by imaging;
4. at least one measurable lesion (according to RECIST v1.1);
5. ECOG score of 0 to 2;
6. expected survival time ≥ 3 months;
7. UGTA1*1*28 and UGTA1*1*6 genes tested wild-type;
8. bone marrow function: neutrophils (ANC) ≥1.5×10^9/L, platelets (PLT) ≥100×10^9/L, hemoglobin (Hb) ≥90g/L, white blood cells (WBC) ≥3.0×10^9/L;
9. Liver function: alanine aminotransferase (ALT), alanine transaminase (AST), alkaline phosphatase (ALP) ≤2.5×ULN (upper limit of normal), ≤5×ULN in case of liver metastasis; total bilirubin ≤1.5×ULN;
10. renal function: serum creatinine (Cr) ≤1.5×ULN or creatinine clearance ≥60 ml/min (calculated according to Cockroft-Gault), urine protein <2+;
11. coagulation: international normalized ratio (INR) ≤ 1.5 times upper limit of normal (ULN) and activated partial thromboplastin time (APTT) ≤ 1.5 times upper limit of normal (ULN);
12. be able to understand the circumstances of this study, and the patient and/or legal representative voluntarily agree to participate in this trial and sign the informed consent form.

Exclusion Criteria:

1. patients who have had other malignant tumors within the previous 5 years (except cured carcinoma in situ and basal cell carcinoma of the skin);
2. prior irinotecan/irinotecan liposome-based chemotherapy;
3. large pleural effusions or ascites requiring intervention;
4. active, uncontrolled bacterial, viral or fungal infections requiring systemic therapy
5. known active HIV infection; untreated active HBV and HCV infection
6. a combination of uncontrolled systemic diseases, including cardiovascular diseases such as unstable angina pectoris, myocardial infarction, congestive heart failure, severe unstable ventricular arrhythmia, and a history of severe pericardial disease; uncontrollable hypertension (defined as systolic blood pressure ≥140 mmHg and/or diastolic blood pressure ≥90 mmHg after regulated antihypertensive medication) or a history of critical hypertension, hypertensive encephalopathy; uncontrollable diabetes; and controlled diabetes mellitus, etc;
7. the presence of severe gastrointestinal-like illness (including active bleeding, greater than grade 1 obstruction, greater than grade 1 diarrhea, or gastrointestinal perforation)
8. history of cesarean section, open thoracic surgery or bowel resection within 28 days prior to enrollment;
9. presence of interstitial pneumonia or pulmonary fibrosis;
10. known hypersensitivity or intolerance to therapeutic drugs or their excipients;
11. history of pulmonary hemorrhage/coughing up ≥ grade 2 (defined as at least 2.5 mL of bright red blood) within 1 month prior to enrollment;
12. presence of arterial embolism, severe hemorrhage (other than hemorrhage due to surgery), or a predisposition to existing embolism or severe hemorrhage within 6 months prior to enrollment
13. presence of central nervous system metastases;
14. the presence of serum albumin ≤ 3 g/dL
15. those using strong inhibitors or inducers of CYP3A4, CYP2C8 and UGT1A1;
16. women who are pregnant or breastfeeding, and patients of childbearing potential who refuse to use adequate contraception during the course of this trial (from study enrollment to the end of primary study focus or surgical treatment);
17. who have participated in another study within 30 days prior to the administration of the first dose of study drug
18. patients who, in the judgment of the investigator, are not suitable for participation in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2025-08-15 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
MPR | After completion of 3 cycle of neoadjuvant therapy (through study completion, an average of half a year)
  Rate of remission of major pathologies

SECONDARY OUTCOMES:
pCR | After completion of 3 cycle of neoadjuvant therapy (through study completion, an average of half a year)
  Pathologic complete remission rate
R0 removal rate | After completion of 3 cycle of neoadjuvant therapy (through study completion, an average of half a year)
  R0 removal rate

IPD SHARING:
Plan to Share IPD: No